CLINICAL TRIAL: NCT02581241
Title: Abnormal QT-Response to the Sudden Tachycardia Provoked by Standing in Individuals With Drug-induced Long QT Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC-15-EC-0379-15-CTIL
Record Dates: First submitted 2015-10-08; First posted 2015-10-20 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Long QT Syndrome
Keywords: QT interval prolongation
MeSH Terms: conditions — Long QT Syndrome | interventions — Tilt-Table Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- drug-induced long QT syndrome (Experimental): 20 adults aged above 18 years which were hospitalized in Tel Aviv medical center between January 2013 and June 2015 due to drug-induced long QT syndrome and the associated torsades de pointes, have no exclusion criteria and provide informed consent to participate in the study.
  Interventions. Participating individuals will be instructed to rest supine for 10 minutes while repeat electrocardiograms are recorded. They will then be instructed to stand up quickly and remain standing still for 10 minutes.
  Individuals with inability to stand up quickly will be tested with tilt table test used in our hospital
  Interventions: Device: tilt table
- control (Active Comparator): 20 adults aged above 18 years which were hospitalized in Tel Aviv medical center between January 2013 and June 2015 and were treated with specific drugs (antibiotics) that potentially prolong the QT interval but they do not have drug-induced long QT syndrome, have no exclusion criteria and provide informed consent to participate in the study.
  Interventions. Participating individuals will be instructed to rest supine for 10 minutes while repeat electrocardiograms are recorded. They will then be instructed to stand up quickly and remain standing still for 10 minutes.
  Individuals with inability to stand up quickly will be tested with tilt table test used in our hospital
  Interventions: Device: tilt table

INTERVENTIONS:
Device: tilt table — Participating individuals will be instructed to rest supine for 10 minutes while repeat electrocardiograms are recorded. They will then be instructed to stand up quickly and remain standing still for 10 minutes.
  Individuals with inability to stand up quickly will be tested with tilt table test used in our hospital

SUMMARY:
The drug-induced long QT syndrome (diLQTS) describes a clinical entity in which administration of a drug produces marked prolongation of the QT interval of the electrocardiogram, associated with the development of a polymorphic ventricular tachycardia, termed torsades de pointes (TdP). The heart rate is an important variable affecting the QT interval. The QT interval normally shortens as the heart rate accelerates; however, the adaptation of the QT interval to sudden heart rate acceleration is not instantaneous. Interestingly, Holter studies show that the speed of response of the QT interval to sudden changes in heart rate (that is, the time it takes the QT interval of a given person to reach a new steady-state QT/RR relation) in healthy persons is highly individual and independent of the basic QTc. The investigators and others recently proposed the "quick standing" test as a simple bedside test that facilitates the diagnosis of congenital LQTS. The test takes advantage of the fact that as one stands up, the heart rate acceleration is abrupt while the associated QT-interval shortening is gradual. As the R-R interval shortens faster than the QT interval, the QT appears to "stretch" toward the next P wave and the corrected QT interval (QTc) for heart rate actually increases momentarily. The phenomenon of "QT stretching" is universal but is exaggerated in patients with LQTS, allowing for a simple but accurate diagnostic test. There is no data on the effects of quick standing on drug-associated form of the long QT syndrome. The investigators therefore propose the present study to better understand who these patients with drug-associated form of the long QT syndrome are and what the significance of their abnormal QT-response is.

DETAILED DESCRIPTION:
The drug-induced long QT syndrome (diLQTS) describes a clinical entity in which administration of a drug produces marked prolongation of the QT interval of the electrocardiogram, associated with the development of a polymorphic ventricular tachycardia, termed torsades de pointes (TdP). Drugs that produce diLQTS block the repolarizing current, IKr, encoded by KCNH2, the disease gene for type 2 congenital LQTS (cLQTS) . Some risk factors are drug-specific (pharmacokinetic factors such as cytochrome P450 variants) whereas others (pharmacodynamic factors) seem more related to myocardial sensitivity across drugs. Studies of the congenital syndrome demonstrated variable penetrance in the congenital syndrome; that is, there is variability in the extent to which mutation carriers display long QT intervals, syncope, and sudden death. Thus, one pharmacogenetic hypothesis is that persons displaying diLQTS represent an atypical form of the congenital form of the syndrome. In fact, a minority of subjects with diLQTS have rare mutations in cLQTS disease genes and can thus be labeled as having the congenital syndrome. In a given family, some persons with a LQTS mutation have clearly long QT intervals, whereas others with the same mutation have normal QT intervals at baseline. In some cases, these latter people, often referred to as "latent" or "subclinical" LQTS, experience TdP only after therapy with a QT-prolonging drug. Indeed, when cLQTS disease genes have been screened, mutations are identified in about 10% of subjects with diLQTS. The heart rate is an important variable affecting the QT interval. The QT interval normally shortens as the heart rate accelerates; however, the adaptation of the QT interval to sudden heart rate acceleration is not instantaneous. Animal and clinical studies have shown that following an abrupt increase in ventricular pacing rate, it takes up to 2 minutes until the ventricular refractory period and the QT interval shorten to a new steady state that is appropriate for the new (faster) rate. Interestingly, Holter studies show that the speed of response of the QT interval to sudden changes in heart rate (that is, the time it takes the QT interval of a given person to reach a new steady-state QT/RR relation) in healthy persons is highly individual and independent of the basic QTc. The investigators and others recently proposed the "quick standing" test as a simple bedside test that facilitates the diagnosis of congenital LQTS. The test takes advantage of the fact that as one stands up, the heart rate acceleration is abrupt while the associated QT-interval shortening is gradual. As the R-R interval shortens faster than the QT interval, the QT appears to "stretch" toward the next P wave and the corrected QT interval (QTc) for heart rate actually increases momentarily. The phenomenon of "QT stretching" is universal but is exaggerated in patients with LQTS, allowing for a simple but accurate diagnostic test. There is no data on the effects of quick standing on drug-associated form of the long QT syndrome. The investigators therefore propose the present study to better understand who these patients with drug-associated form of the long QT syndrome are and what the significance of their abnormal QT-response is.

ELIGIBILITY:
Inclusion Criteria:

* age above 18 years
* were hospitalized in Tel Aviv medical center between January 2013 and June 2015 due to drug-induced long QT syndrome and the associated torsades de
* were treated with specific drugs (antibiotics) that potentially prolong the QT interval (only for control group)

Exclusion Criteria:

* Subjects with an inability to communicate well with the investigators (i.e., language problem, poor mental development or impaired cerebral function).
* Subjects with any acute medical situation (e.g. acute infection) within 48 hours of study start, which is considered of significance by Investigator.
* Subjects who are non-cooperative or unwilling to sign consent form.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-08-17 (Actual); Study Completion 2017-08-23 (Actual)

PRIMARY OUTCOMES:
ECG measurements of QT before and during stand up test | 12 months
  ECG measurements of QT and RR before and during stand up test. measured in msec units

CONTACTS AND LOCATIONS:
Overall Officials: Udi Chorin, MD, Principal Investigator — Tel Aviv MC
Locations (1):
- Sourasky medical center (Ichilov), Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No